CLINICAL TRIAL: NCT01539486
Title: Relationship of Preoperative PTH and Ex-Vivo Gamma Counts in Minimally Invasive Parathyroidectomy
Brief Title: Relationship of Preoperative Parathyroid Hormone (PTH) and Ex-Vivo Gamma Counts in Minimally Invasive Parathyroidectomy
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 112684
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-01

CONDITIONS: Parathyroid Disease
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The intent for this study is to do a retrospective chart review of all patients who have undergone minimally invasive parathyroidectomy for primary hyperthyroidism. All data collected will be recorded under assigned identification numbers that will have no association with medical record or hospital numbers. Identifying characteristics will include age and sex. Anonymity will be upheld. The patient/family will not be contacted directly. All information will be obtained from the medical chart. Demographics, location, preoperative PTH levels and intraoperative Ex-Vivo gamma counts, co-morbid conditions, and the outcome based on the hospital notes will be obtained from patients' charts and will be transferred to a secure database. It is our hypothesis that there is a linear relationship between immediate preoperative parathyroid hormone (PTH) levels and Ex-Vivo gamma counts and the aim of this study is to better describe this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between the ages of 18 and 90 years old who have documented primary hyperparathyroidism and have undergone minimally invasive parathyroidectomy.

Exclusion Criteria:

* Patients who have not had both intraoperative parathyroid hormone (PTH) levels and Gamma counts during their parathyroidectomy
* Patients who have parathyroidectomies for reasons other than primary hyperparathyroidism.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An estimated 200 patient charts will be reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2010-01; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Retrospective Chart Review | Retrospective Chart Review
  The information presented in this report will provide a surgical tool for otolaryngologists to improve the efficiency and efficacy in patients with hyperparathyroid disease.

CONTACTS AND LOCATIONS:
Overall Officials: Deanne King, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States